CLINICAL TRIAL: NCT04424576
Title: Trajectory of Ovarian Morphology During the Adolescent Reproductive Transition
Brief Title: Ovarian Morphology in Girls
Acronym: OMG
Status: Recruiting | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 0000779
Record Dates: First submitted 2020-05-18; First posted 2020-06-11 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Amenorrhea; Oligomenorrhea; Puberty
Keywords: Ovary; Transabdominal Ultrasound; Menarche; Periods; Microbiome
MeSH Terms: conditions — Amenorrhea; Oligomenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular Menstrual Cycles: 22 adolescents with regular menstrual cycles (i.e., once every 4-6 weeks) will be enrolled within 11 months of menarche.
- Irregular Menstrual Cycles: 26 adolescents with irregular menstrual cycles (i.e., < 4 weeks or > 6 weeks between periods) will be enrolled within 11 months of menarche.

SUMMARY:
Establishment of regular menstrual cycles is a key component of reproductive maturation and a recognized vital sign for health and well-being. Irregular menstrual cycles are especially common for the first 2-3 years after an adolescent's first menstrual period (i.e., menarche), which delays the identification and diagnosis of early reproductive disturbances such as polycystic ovary syndrome (PCOS). The purpose of this research study is to determine whether the ovary can serve as a reliable predictor of normal or abnormal development by following the trajectory of ovarian morphology in conjunction with menstrual cyclicity using 3D transabdominal ultrasound imaging in a prospective cohort study of adolescents. A secondary objective is to identify potential environmental factors such as diet and the gut microbiome which influence the trajectory towards normal or abnormal reproductive development.

DETAILED DESCRIPTION:
Establishment of regular menstrual cycles is a key component of reproductive maturation and a recognized vital sign for health and well-being. Irregular menstrual cycles are especially common for the first 2-3 years after an adolescent's first menstrual period (i.e., menarche), which delays the identification and diagnosis of early reproductive perturbations and subsequent future disease risk. Therefore, the objectives of this study are to determine whether there are distinct aspects of ovarian morphology that predict the likelihood of regular menses or cycle irregularity at 2y post-menarche and to determine whether diet or lifestyle (such as quality of sleep) contribute to changes in the ovaries and period patterns.

A group of up to 60 adolescents will be enrolled into a prospective longitudinal cohort study. Participants will attend four study visits to their location's respective clinical research center. Study visits will occur at four distinct time points post-menarche: 6-10 months, 11-13 months, 17-19 months, and 23-25 months.

Prior to each of the study visits, participants will undergo one planned 24-hr dietary recall by a member of the research team and self-collect a stool sample.* Participants will be asked to fast the night before the study visit. At each study visit, participants will undergo the following assessments:

A 3D transabdominal ultrasound of the ovaries and uterus.

A fasting blood sample, obtained via venipuncture.

A series of anthropometric assessments, including: height, weight, waist and hip circumference, blood pressure, heart rate, and body fat percentage obtained using a bioimpedance scale.

Tanner stage assessment, using a standardized self-report scoring scheme and by a trained member of the research team who is blinded to the results of the self-reported tanner stage.

Acne scoring, using a standardized scoring scheme by a member of the research team.

Hirsutism assessment, obtained by visually inspecting nine pre-defined regions of the body for terminal hair growth using a standardized scoring scheme by a trained member of the research team.

Urine sample, self-collected by the participant after the transabdominal ultrasound.*

24-hour dietary recall.*

Physical activity questionnaire.*

Two sleep questionnaires, including questions about sleep hygiene, sleep quality, and circadian rhythms.*

In between study visits, participants will maintain menstrual cycle diaries and medication diaries.

*Participants at the University of Rochester site will not complete the urine or stool collection, the dietary recalls, or any of the physical activity and sleep questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents aged 9 to 17 years
* Menarche within 11 months of the enrollment visit
* University of Rochester site only: Family history of PCOS (i.e., mother or aunt)

Exclusion Criteria:

* Current or recent use of medications or supplements known or suspected to interfere with reproductive or metabolic function in the past 2 months (e.g., contraceptives, metformin, steroids, anti-seizure medications)
* Untreated and/or unstable medical or mental health condition known or suspected to interfere with reproductive or metabolic function
* Currently pregnant or breast feeding
* History of ovarian surgery
* Presence of significant acute or chronic illness which may interfere with study participation

Ages: 9 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Eligibility is limited to biologically female individuals because the primary study endpoints include the ovary and menstrual cycle.
Study Population: Female adolescents between the ages of 9 and 17 years who achieved menarche (i.e., very first period) within the past 11 months will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Ovarian size | 24 months
  Changes in ovarian size over the first 2y post-menarche will be assessed and compared across cohorts.
Follicle counts | 24 months
  Follicle counts, expressed as follicle number per ovary (FNPO) and follicle number per cross-section (FNPS), will be assessed over the first 2y post-menarche and compared across cohorts. Numbers of large follicles (>10 mm diameter) and small follicles (<10 mm diameter) will also be compared across cohorts.
Menstrual cycle status | 24 months
  Menstrual cycle status (i.e., regular versus irregular menstrual cycles) will be assessed using menstrual cycle records maintained by participants over the course of the study. Changes in menstrual cycle status over the 2y post-menarche and relationships between menstrual cycle status and other physiological and lifestyle factors will be examined.

SECONDARY OUTCOMES:
Body composition | 24 months
  Changes in percent body fat, obtained using a bioimpedence scale, will be assessed over the first 2y post-menarche and compared across cohorts.
Leutenizing hormone (LH), follicle stimulating hormone (FSH), estradiol, progesterone, anti-mullerian hormone, free and total testosterone, and androstenedione | 24 months
  Serum levels of these reproductive hormones will be assessed over the first 2y post-menarche and compared across cohorts.
Sleep quality | 24 months
  Sleep quality will be assessed using two questionnaires: the Morningness-Eveningness Scale for Children and the Children's Report of Sleep Patterns. Sleep quality will be assessed over the first 2y post-menarche and compared across cohorts.
Dietary composition | 24 months
  Dietary composition (i.e., macro and micronutrient totals, total energy intake) will be assessed using two 24-Hour Food Frequency Questionnaires administered at each gynecological time point.
Gut microbiome richness and diversity | 24 months
  Gut microbiome richness and diversity will be assessed over the first 2y post-menarche and compared across cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Marla E Lujan, PhD, Principal Investigator — Cornell University; Tania Burgert, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Romina Barral, MD MSCR FAPP, Principal Investigator — Children's Mercy Hospital Kansas City; Kathleen Hoeger, MD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cornell University - Human Metabolic Research Unit, Ithaca, New York
  - University of Rochester, Strong Fertility Center, Rochester, New York